CLINICAL TRIAL: NCT00342576
Title: Host Response to Infection and Treatment in Lymphatic Filarial Disease Strongyloidiasis in India
Brief Title: Host Response to Infection and Treatment in Lymphatic Filarial Disease in India
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 9999890048; OH89-I-0048
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07-15

CONDITIONS: Lymphatic Filarial Disease
Keywords: Filarial Parasites; Wuchereria Bancrofti; Brugia Malayi; Diethylcarbamazine (DEC); Ivermectin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Patients admitted on this protocol will have, or be suspected of having, one of the lymphatic filarial infections affecting humans. After routine clinical evaluation they will be studied in depth immunologically, and their blood cells and/or serum will be collected to provide reagents (eg., specific antibodies, T cell clones, etc.) that will be used in the laboratory to address the broader questions of immunodiagnosis, immunoregulation, immunopathology and immunoprophylaxis. Careful observations of the patients' clinical and immunologic responses to therapy will be made, as well as long-term follow-up of these changes. It is anticipated both that the patients will receive optimal clinical care for their infections and that the specimens collected from them will prove to be valuable reagents for the laboratory studies of the immunologic responses unique to filarial or other helminthic infections.

DETAILED DESCRIPTION:
This study is designed to determine the presence of and the immune response to filarial and stronglyloides infections in an area endemic for both infections in South India. This study will aim to examine the presence of filarial and Strongyloides stercoralis infection at a community level as well as in hospital settings. After routine clinical evaluation and screening, individuals enrolled in this protocol will be studied in depth immunologically, and their blood cells and/or serum will be collected to address the broader questions of immunodiagnosis, immunoregulation and immunopathology. Careful observations of the individual s clinical and immunologic responses to therapy will be made, as well as long-term follow-up of these changes. In addition to infected individuals, this protocol will also be used to study individuals with filarial pathology and endemic normal individuals. This will enable us to characterize the immunological profiles of infected, uninfected and diseased individuals in an endemic area and provide greater insight into the pathogenesis of lymphatic filarial disease as well as the immunology of strongyloides infection.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 18-75 years.

Ability to give informed consent.

EXCLUSION CRITERIA:

Pregnant or nursing women will be excluded from the treatment arm of the study.

Less than 18 years of age; greater than 75 years of age.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 1994-04-23; Study Completion 2019-07-15

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Nutman, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Tuberculosis Research Centre, Chennai, India

REFERENCES:
- [Background] Piessens WF, Partono F, Hoffman SL, Ratiwayanto S, Piessens PW, Palmieri JR, Koiman I, Dennis DT, Carney WP. Antigen-specific suppressor T lymphocytes in human lymphatic filariasis. N Engl J Med. 1982 Jul 15;307(3):144-8. doi: 10.1056/NEJM198207153070302. PMID 6178026
- [Background] Nutman TB, Kumaraswami V, Pao L, Narayanan PR, Ottesen EA. An analysis of in vitro B cell immune responsiveness in human lymphatic filariasis. J Immunol. 1987 Jun 1;138(11):3954-9. PMID 3295043
- [Background] Nutman TB, Kumaraswami V, Ottesen EA. Parasite-specific anergy in human filariasis. Insights after analysis of parasite antigen-driven lymphokine production. J Clin Invest. 1987 May;79(5):1516-23. doi: 10.1172/JCI112982. PMID 3553242